CLINICAL TRIAL: NCT07099924
Title: Bilateral Rectus Sheath Catheters Following Midline Laparotomy. A Randomized, Placebo-controlled Trial
Brief Title: Rectus Sheath Catheters Following Midline Laparotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepios Kliniken Hamburg GmbH (Other)
Responsible Party: Principal Investigator, Ronald Seidel, Head of Anesthesia and Intensive Care, Asklepios Kliniken Hamburg GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-87-BO-ff
Record Dates: First submitted 2025-07-16; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acute Abdomen; Ileus; Colorectal Carcinoma
Keywords: postoperative analgesia; rectus sheath catheter; ultrasound; midline laparotomy
MeSH Terms: conditions — Abdomen, Acute; Ileus; Colorectal Neoplasms | interventions — Anesthetics, Local; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: single center, randomized, placebo-controlled, observer-blinded
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ropivacaine 0.2% (Experimental): 2x30 ml (bilateral) ropivacaine 0.2% every 8 hours
  Interventions: Drug: Ropivacaine 0.2%
- saline 0.9% (Placebo Comparator): 2x30 ml (bilateral) saline 0.9% every 8 hours
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Ropivacaine 0.2% — 2x30ml (bilateral) ropivacaine 0.2% every 8 hours via rectus sheath catheter
  Other Names: local anesthetic
  Arms: ropivacaine 0.2%
Drug: Saline 0.9% — 2x30ml saline 0.9% every 8 hours via rectus sheath catheter
  Other Names: placebo
  Arms: saline 0.9%

SUMMARY:
Rectus sheath catheters (RSC) are used for postoperative analgesia following midline laparotomies. Local anesthetics are applied to the posterior rectus sheath via the RSC. The target structures are the anterior cutaneous branches of the spinal nerves Th7-Th12. RSC can be used in particular if thoracic epidurals are contraindicated (compromised coagulation), technically unfeasible or refused by the patient.

The study investigates placebo-controlled weather RSC have a significant additional analgesic effect in a multimodal analgesic concept. Primary outcome parameters are the maximum pain score, the Quality-of-Recovery-15-Score (QoR-15GE) and the opioid consumption (morphine equivalents) in the first 72h postoperatively.

DETAILED DESCRIPTION:
Recruitment Patients are recruited during the anesthesiology consultation. Patients who provided written informed consent. fulfill all inclusion and no exclusion criteria will be included in the study.

Allocation of study medication After inclusion in the study, each patient receives a patient number, which is noted on the Case Report Form (CRF). The randomization list was generated via www.random.org (Randomness and Integrity Services Ltd., Dublin, Ireland). Random assignment to groups 1 (verum) and 2 (placebo) was performed on the day of surgery using the sealed envelope technique. The sealed envelope is opened by a doctor not involved in the study immediately before bilateral placement of the rectus catheters catheters. This colleague prepares the study medication (verum or placebo, unlabeled, blinded to the observer and patient).

Anesthesia and perioperative monitoring After a peripheral or central venous line is inserted, a balanced electrolyte solution is connected and the following parameters are monitored until complete postoperative recovery: blood pressure (plethsymographic or via arterial line), electrocardiogram, pulse oximetry.

The surgical procedures are performed under general anesthesia (sevoflurane 0.7-1.0 MAC). Sufentanil (0.2-0.4 microg/kg), propofol (1.5-2 mg/kg) and cisatracurium (0.1-0.15 mg/kg) are administered to induce anesthesia The multimodal analgesia concept includes the intraoperative administration of 4 mg dexamethasone (antiemetic, coanalgesic) and two non-opioids: 1 g metamizole (40 mg parecoxib if contraindications exist) and 1 g paracetamol.

Study intervention Bilateral RSC are placed intraoperatively after closure of the median laparotomy under aseptic conditions, before the wound dressing is applied. For imaging, we use an ultrasound device (FUJIFILM Sonosite, Bothel, WA, USA) with a linear transducer (38mm, 6-13MHz), which is placed obliquely on the upper edge of the median laparotomy. The puncture (puncture direction from medial-cranial to lateral-caudal) is initially performed with an ultrasound-optimized single-shot cannula (SonoPlex 22G50mm to 21G100mm, Pajunk, Geisingen, Germany) in order to reliably identify the compartment of the posterior rectus sheath. After verification of the correct spread of the local anesthetic, the catheter (SonoLong Echo 19G 50-100mm, 20G 50cm catheter, Pajunk, Geisingen, Germany) is placed at the lateral edge of the posterior rectus sheath and again the correct spread of the local anesthetic in the target compartment is verified by ultrasound.

Group 1 Verum (ropivacaine 0.2%) Dosage 2x30ml ropivacaine 0.2% every 8h (120mg every 8h) Daily dose 360mg

Group 2 Placebo (saline 0.9%) Dosage 2x30ml saline 0.9% every 8h

Postoperative care Postoperatively, patients are cared for in the recovery room or intensive care unit. As soon as their condition allows, they are transferred to a peripheral ward. Non-opioid analgesics are continued. An additional opioid-based on-demand medication is prescribed (7.5 mg piritramid), the dose of which is documented as morphine equivalents (5 mg).

ELIGIBILITY:
Inclusion Criteria:

* Median laparotomy
* Age over 18 years
* Informed consent has been obtained

Exclusion Criteria:

* Local signs of inflammation
* known allergy to local anesthetics used
* chronic pain syndrome
* drug addiction
* post-operative ventilation that cannot be completed on the day of surgery
* lack of consent or cooperation
* pregnancy
* participation in another medical study
* sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | on first postoperative day
  Quality-of-Recovery Score 15, minimum value 0, maximum value 150, higher values mean a better outcome
pain score (numeric rating scale) | daily up to 72 hours postoperatively
  at rest and at movement, minimum value 0, maximum value 10, lower values mean a better outcome
Opioid consumption | on the day of surgery, on the first postoperative day, on the second postoperative day, on the third postoperative day
  cumulative morphine equivalents

SECONDARY OUTCOMES:
postoperative complications | up to 14 days from date of randomization
  Number of participants experiencing the following postoperative complications:
  nausea and vomiting, constipation, respiratory failure, pneumonia, wound infections, wound dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Seidel, Dr.med., Principal Investigator — Asklepios Klinikum Uckermark
Locations (1):
- Asklepios Medical Center Uckermark, Schwedt, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: up to 6 months after publication
Access Criteria: on request to the principal investigator